CLINICAL TRIAL: NCT05175924
Title: The Effect of Virtual Reality On Pain and Anxiety During Blood Draw in Children: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Gülsün Ayran, Asistant Professor, Erzincan Binali Yildirim Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Erzi̇ncanBinaliYildırim
Record Dates: First submitted 2021-10-26; First posted 2022-01-04 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Pain, Procedural; Children, Only
Keywords: Anxiety; Blood draw; Children; Nursing; Pain; Virtual reality
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial consisting of an experiment and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental): In the Aquarium VR group, virtual reality headset compatible with iPhone 7 (Apple) was used to distract attention. Before use, the headsets were tested on five children for face fit and visibility of the application used. Written and verbal consent of the children and their parents was obtained to test the headsets. The children who tested the headsets were not included into the study. The headset offered a soft and comfortable experience in contact with the skin due to its leather and pad covering. It also had a wide viewing angle and an optical zoom button. Due to its noise isolation function, it did not disturb anyone or make noise.
  Interventions: Other: Nanpharmacological method

INTERVENTIONS:
Other: Nanpharmacological method — Virtual Reality

SUMMARY:
Purpose: The study was carried out to determine the effect of virtual reality applied during blood collection upon pain and anxiety in children aged 5-12.

Design and Methods: In this randomized controlled study, children included in the sample group were assigned to the control group (n=43) and Aquarium VR group (n=45) using block randomization. "Child State Anxiety Scale " and "Wong-Baker Faces Pain Scale" were used to collect the data of the study. Children in the Aquarium VR group watched the "Aquarium VR" application through virtual reality glasses during the procedure. The children in the control group benefited from routine nursing services. The pain scores after blood collection and anxiety scores before and during blood collection in children in both groups were interpreted.

DETAILED DESCRIPTION:
Purpose: The study was carried out to determine the effect of virtual reality applied during blood collection upon pain and anxiety in children aged 5-12.

MATERIAL AND METHOD Study Design, Participants This study in randomized controlled design was carried out with children aged between 5-12 in Pediatric Polyclinic blood draw unit of the University Hospital in a province in Turkey between 15 May and 31 July 2021. The study population included children who applied to the Pediatrics Polyclinic blood draw unit of the prespecified hospital between 15 May-31 July 2021. It was calculated by taking into account the pre-test anxiety score averages of the intervention and control groups in the study of Gerker et al. (2019) (for the t-test to compare the two groups). As a result of the evaluations, it was calculated as d=0.99 (high effect size), power=0.95, α=0.05 in the G*Power 3.1.9.2 statistical program. Accordingly, it was determined that the minimum number of children to be included in the study was 28 for the intervention group and 28 for the control group, a total of 56 children. Between these dates, 45 patients were included in the experimental group and 43 patients in the control group, who met the research criteria and volunteered to participate in the research, and the study was completed with a total of 88 patients. The study was carried out with children aged 5-12 years, who did not have communication barriers, did not use glasses, did not have pain before the procedure and did not have a chronic disease that would cause pain, blood was taken from the antecubital region and volunteered to participate in the study.

Randomization The children were included in groups randomly. "Stratification and block randomization methods" were used in the study for assigning the participants to the control and study groups. It was reported in the literature that the variables of age, gender, and interventional procedure experience were among the factors affecting the pain and anxiety experienced by children during interventional procedures. In this sense, the children were stratified as "female and male" for the gender variable and "5-8 years and 9-12 years" for the age variable, and block randomization was performed. In order to prevent the groups from being influenced by each other, data of the study group were collected in one day and the control group in the other. Data collection days of the study and control groups were determined with the method of drawing lots. This cycle was continued until sufficient sample size was obtained.

Data Collection Tools Question Form In this section, there were 6 questions related to the descriptive characteristics of the children (age, gender, education level of the mother, education level of the father, time of the last blood draw, the parent's presence with the child during the blood draw process).

Wong Baker Faces Pain Scale-WBFPS This scale measuring the severity of pain was used in children aged between 3-18 years. In this scale, pain was scored for facial expressions according to numerical values, and the numerical rating of the scale varied between 0 and 10. Facial expressions ranging from smiling (0=very happy/no pain) to crying (10=most painful) indicated emotions. The severity of pain increased as the score obtained from the scale increased, and the severity decreased as the score decreased. The child was possible to tell the nurse about the pain experienced more accurately with the drawing illustrating what each of the different numbers on the pain scale indicated. This scale was a reliable measurement tool for the Turkish population (Tsao and Zeltzer, 2008).

Children's State Anxiety Scale (CSAS) CSAS was a thermometer-like scale with a light bulb at the bottom and horizontal upward lines at intervals. On the scale, the children were instructed as "Imagine all your anxious or frustrated feelings are in the bulb or bottom of the thermometer." "If you're a little worried or nervous, emotions can go a little upward on the thermometer. If you are very, very anxious or nervous, the emotions can go to the top. Put a line indicating how worried or angry you are on the thermometer." In order to measure state anxiety (CSAS), the children were asked to mark what they felt "right now". Before filling in CSAS, sequencing skills of the children were monitored. They were asked to count to ten, They were also asked to answer, "Which is bigger, seven or four?" The children who could not successfully complete these tasks or did not understand the instructions were not asked to fill in CSAS. Subsequent to data collection, two members of the research team reviewed and scored CSAS of the children. A transparent meter with increments of ½ point marked was placed above the rating of children, then the increment of ½ point was rounded to the nearest number. The score varied between 0 and 10 (Gerçeker et al., 2018).

Virtual Reality Headset In the Aquarium VR group, virtual reality headset compatible with iPhone 7 (Apple) was used to distract attention. Before use, the headsets were tested on five children for face fit and visibility of the application used. Written and verbal consent of the children and their parents was obtained to test the headsets. The children who tested the headsets were not included into the study. The headset offered a soft and comfortable experience in contact with the skin due to its leather and pad covering. It also had a wide viewing angle and an optical zoom button. Due to its noise isolation function, it did not disturb anyone or make noise.

"Aquarium VR" Application The application simulated a submarine journey to explore the inside of virtual aquarium. The aquarium included sharks, aquatic mammals, clown fish and much more. It also allowed children to learn more about marine life in the Pacific Ocean (Eon Reality, 2021).

Ethical Principles of the Research In order to carry out the research, 14/03/2021 dated and 03/14 numbered ethics committee approval from the Human Research Ethics Committee and legal permissions from the Hospital Management were obtained. After informing the children participating in the study and their parents about the research, they were explained about being free to participate in or not, and their written and verbal consent was also obtained from the parents. The children who participated into the study and their parents were assured that their personal information would not be disclosed to others, would not be used anywhere else and they had right to withdraw from the study at any time they wanted.

Data Collection The children included into the study and control groups and their families were primarily informed about the study by the researcher in the waiting room at the entrance of the pediatric outpatient clinic blood draw unit. The children who were in 5-12 age group, had no communication barriers, did not use glasses, had no pain before the procedure and did not have a chronic disease causing pain, and volunteered to participate into the study were included in the study. The "Informed Consent Form" was signed by the parents and children who met the criteria and agreed to participate into the study. The children were stratified as "female and male" for the gender variable and "5-8 years and 9-12 years" for the age variable, and block randomization was performed.

The children included into the study and control groups and their parents were asked to rate CSAS to assess their anxiety levels before and during blood draw, and WBFPS to determine the pain they felt in their arm during blood draw. Similarly, the nurse and researcher rated WBFPS and CSAS.

The children in the study group were shortly informed about using the virtual reality glasses before the procedure. When the children sat on the patient's chair for blood draw, they put on virtual reality glasses and 3D "Aquarium VR" application was started to be watched from the virtual reality glasses 1 minute before the blood draw procedure. At the same time, the nurse applied a tourniquet for blood draw from the child and determined the vein from which blood would be drawn from the antecubital region. The blood was drawn from the antecubital region by the same nurse by means of a vacuum blood draw tube and the process lasted for approximately 2-3 minutes. During this procedure, the children were asked not to remove their virtual reality glasses at all.

No interventional procedure was administered to the children in the control group. Blood was drawn from the antecubital region by the same nurse by means of a vacutainer. In both groups, parents were permitted to be with their children in the blood draw room during the procedure.

Data Analysis and Interpretation SPSS 25.0 package software was used for statistical analysis of the data. Percentage, average, Simple t-test and One Way ANOVA analysis were used to interpret the data. The statistical level of significance was regarded to be 0.05 in all tests. In order to obtain statistical results, fit of the data to the normal distribution was interpreted using the Shao method. In this sense, the Skewness value was determined to be 0.139, the Kurtosis value was -2,027, and it was found to have a normal distribution between -3 and +3.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 5-12 years old
* There should be no pain before the blood draw procedure
* Should not have a chronic disease that will cause pain Blood should be taken from the antecubital region
* Must be willing to participate in the research

Exclusion Criteria:

* The transmission barrier
* Wearing glasses
* Involuntary

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Wong-Baker Faces Pain Scale Mean Scores by Groups | Evaluated at the time of blood collection.
  This scale measuring the severity of pain was used in children aged between 3-18 years. In this scale, pain was scored for facial expressions according to numerical values, and the numerical rating of the scale varied between 0 and 10. Facial expressions ranging from smiling (0=very happy/no pain) to crying (10=most painful) indicated emotions.

SECONDARY OUTCOMES:
Comparison of Child Anxiety Scale Mean Scores before and during the procedure according to the groups | Evaluated before and during blood collection.
  CSAS was a thermometer-like scale with a light bulb at the bottom and horizontal upward lines at intervals. On the scale, the children were instructed as "Imagine all your anxious or frustrated feelings are in the bulb or bottom of the thermometer." "If you're a little worried or nervous, emotions can go a little upward on the thermometer. If you are very, very anxious or nervous, the emotions can go to the top. Put a line indicating how worried or angry you are on the thermometer." A transparent meter with increments of ½ point marked was placed above the rating of children, then the increment of ½ point was rounded to the nearest number. The score varied between 0 and 10

CONTACTS AND LOCATIONS:
Locations (1):
- Gülsün Ayran, Merkez, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No